CLINICAL TRIAL: NCT03475212
Title: Antiviral Cellular Therapy for Enhancing T-cell Reconstitution Before or After Hematopoietic Stem Cell Transplantation (ACES) PBMTC SUP1701
Brief Title: Antiviral Cellular Therapy for Enhancing T-cell Reconstitution Before or After Hematopoietic Stem Cell Transplantation
Acronym: ACES
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pediatric Transplantation & Cellular Therapy Consortium (Other)
Responsible Party: Principal Investigator, Michael Pulsipher, Sponsor-Investigator, Protocol Co-Chair, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBMTC SUP1701
Record Dates: First submitted 2018-01-13; First posted 2018-03-23 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-03

CONDITIONS: Cytomegalovirus Infections; Adenovirus Infection; EBV Infection
Keywords: Hematopoietic Stem Cell Transplant; Primary Immune Deficiency Disease
MeSH Terms: conditions — Cytomegalovirus Infections; Adenoviridae Infections; Epstein-Barr Virus Infections; Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virus specific T cell lines (VSTs) against three viruses (Experimental): The study will evaluate whether partially-HLA matched allogeneic multivirus-specific VSTs, activated using overlapping peptide libraries spanning immunogenic antigens from CMV, adenovirus and EBV, will be safe and produce anti-viral effects in immunodeficient recipients infected with one of more of the targeted viruses that are persistent despite conventional anti-viral therapy.
  Interventions: Biological: Virus Specific T-cell (VST) infusion

INTERVENTIONS:
Biological: Virus Specific T-cell (VST) infusion — Patients will receive partially HLA-matched VSTs as a single infusion. Patients who have a partial response (>1 log decrease in viral load without clearance) or no response and do not have treatment-related dose-limiting toxicities are eligible to receive up to 3 additional doses from day 30 after the initial infusion and at 2 weekly intervals thereafter. The viral load of the virus (or viruses) that patients are initially treated for are monitored by viral PCR.

SUMMARY:
The purpose of this study is to evaluate whether virus-specific T cell lines (VSTs) are safe and can effectively control three viruses (EBV, CMV, and adenovirus) in patients who have had a stem cell transplant and also in patients that have a primary immunodeficiency disorder with no prior stem cell transplant.

DETAILED DESCRIPTION:
The primary purpose of the study is to evaluate whether most closely HLA-matched multivirus-specific T cell lines obtained from a bank of allogeneic virus-specific T cell lines (VSTs) have antiviral activity against three viruses: EBV, CMV and adenovirus.

Reconstitution of anti-viral immunity by donor-derived VSTs has shown promise in preventing and treating infections associated with CMV, EBV and adenovirus post-transplant. However, the time required to prepare patient-specific products and lack of virus-specific memory T cells in cord blood and seronegative donors, limits their value. An alternative is to use banked partially HLA-matched allogeneic VSTs. A prior phase II study at Baylor College of Medicine using trivirus-specific VSTs generated using monocytes and EBV-transformed B cells gene-modified with a clinical grade adenoviral vector expressing CMV-pp65 to activate and expand specific T cells showed the feasibility, safety and activity of this approach for the treatment of refractory CMV, EBV and Adenovirus infections. More recent protocols utilizing synthetic viral peptide pools allow ex vivo expansion of T-cells targeting multiple viral antigens in 10-12 days without use of viral transduction.

The study will evaluate whether partially-HLA matched allogeneic multivirus-specific VSTs, activated using overlapping peptide libraries spanning immunogenic antigens from CMV, adenovirus and EBV, will be safe and produce anti-viral effects in immunodeficient recipients infected with one of more of the targeted viruses that are persistent despite conventional anti-viral therapy.

This study will evaluate safety and efficacy of partially-matched VST therapy in A) patients who have persistent viral infections in the post-HSCT period, and B) patients with primary immunodeficiency conditions who have persistent viral infections and have not undergone HSCT.

The study agent will be assessed for safety and antiviral activity.

ELIGIBILITY:
Inclusion Criteria

Patients who have received any type of allogeneic transplant or who have a primary immunodeficiency disorder will be eligible if they have CMV, adenovirus, and/or EBV infection/disease with failure of treatment after 7 days of standard therapy OR if unable to tolerate standard therapy.

* Patients must meet one of the following criteria:

  * Recipient of prior myeloablative or non-myeloablative allogeneic hematopoietic stem cell transplant using either bone marrow or peripheral blood stem cell or single or double cord blood within the previous 18 months, OR
  * Have a diagnosed primary immunodeficiency disorder (as defined by clinical and laboratory evaluations) and not undergone HSCT.
* Treatment of the following persistent or relapsed infections despite standard therapy:

  * CMV: Treatment of persistent or relapsed CMV disease or infection after standard therapy. For CMV infection, standard therapy is defined as antiviral therapy with ganciclovir, foscarnet or cidofovir for at least 14 days.
  * Adenovirus: Treatment of persistent or relapsed adenovirus infection or disease despite standard therapy. Standard therapy is defined as antiviral therapy with cidofovir or brincidofovir.
  * EBV: Treatment of persistent or relapsed EBV infection despite standard therapy.

For EBV infection, standard therapy is defined as rituximab given at 375 mg/m2 in patients for 1-4 doses with a CD20+ tumor.

Additional Inclusion Criteria:

* Patients with simultaneous infections with CMV, EBV and/or Adenovirus infections are eligible if one or more infection(s) is persistent or relapsed despite standard therapy as defined above. Patients with multiple infections with one or more reactivation and one or more controlled infection are eligible to enroll.
* Clinical status at enrollment that allows tapering of steroids to equal or less than 0.5 mg/kg/day prednisone (or equivalent) prior to infusion of the VST doses.
* Negative pregnancy test in female patients if applicable (childbearing potential who have received a reduced intensity conditioning regimen).
* Written informed consent and/or signed assent line from patient, parent or guardian.

Exclusion Criteria

* Patients receiving ATG, Campath, Basiliximab or other immunosuppressive monoclonal antibodies targeting T-cells within 28 days of screening for enrollment.
* Patients who have received donor lymphocyte infusion (DLI) or other experimental cellular therapies within 28 days.
* Current therapy with ruxolitinib or other JAK inhibitors within the previous 3 days.
* Patients with other uncontrolled infections, defined as bacterial or fungal infections with clinical signs of worsening despite standard therapy. For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment. For fungal infections, patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to enrollment.
* Progressing infection is defined as hemodynamic instability, worsening physical signs, or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
* Patients with active and uncontrolled relapse of malignancy (if applicable).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility to identify suitable HLA matched VST products | 30 days
  Feasibility will be defined as the ability of the investigators to identify suitable partially HLA- matched VST products from the VST bank at Children's National Medical Center for referred study subjects. The percentage of referred patients with potential partially-matched VST products identified will be recorded, as will timing between patient referral and treatment.
Incidence of Treatment-Emergent Adverse Events | 30 days
  The safety endpoint, dose-limiting toxicity (DLT), will be defined as acute GvHD grades III-IV or grades 3-5 infusion-related adverse events or grades 4-5 non-hematological adverse events related to the T cell product within 30 days of each VST dose and that are not due to the pre-existing infection or the original malignancy or pre-existing co-morbidities as defined by the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03.
Efficacy of VST at 30 days as measured by viral load | 30 days
  Peripheral blood and, where relevant, stool and urine will be monitored for CMV, EBV, and/or adenovirus viral load. For patients with multiple viral infections, the response against the primary viral target will determine the classification. For the infection under treatment response in viral load will be assessed at 30 days after the first VST infusion

SECONDARY OUTCOMES:
Reconstitution of Antiviral Immunity following VST infusions | 3 months
  Patient serum and peripheral blood mononuclear cells will be monitored for virus-specific activity during the 3 months following VST infusion by the following measures:
  1. T cell phenotyping by flow cytometry (including % CD3, CD4, CD8, TCRalpha/beta and CD45RA-/CCR7+, among other markers)
  2. Antiviral T cell responses to CMV, EBV, and/or Adenovirus antigens by IGN-g ELIspot (spot forming units) and Intracellular cytokine staining ( %IFN-gamma and TFNa+ of CD4 and CD8 cells)
  3. T cell repertoire and antiviral specificity by TCR sequencing (%clonotype frequencies)
Persistence of infused VSTs | 1 month and 3 months
  Persistence of infused T cells will be monitored at 1 month and 3 months following VST infusion using deep sequencing and additional tests as indicated to track the TCR v-beta repertoire in the patient peripheral blood prior to and post-infusion.
Effects on Clinical Signs of Viral Infection | 3 months
  If a patient has organ involvement, clinical response will be monitored. For patients with EBV lymphoma and measurable disease, response will be assessed by RECIST criteria.
Survival | 6 months and 12 months
  Overall survival at 6 and 12 months post VST infusion will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pulsipher, MD, Study Chair — Children's Hospital Los Angeles; Michael Keller, MD, Study Chair — Children's National Research Institute
Locations (30):
- United States (30):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - City of Hope, Duarte, California
  - University of California, Los Angeles, Los Angeles, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford Lucile Packard Children's Hospital, Palo Alto, California
  - UCSF Medical Center, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Emory University/Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children - Indiana University, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute/ Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Spectrum Health - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - The Children's Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Jude, Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Children's Mercy, San Antonio, Texas
  - Methodist Healthcare System of San Antonio, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center/Seattle Chlindren's/University of Washington School of Medicine, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No